CLINICAL TRIAL: NCT04171687
Title: A Randomized, Open-label, Multiple-dose, Crossover Clinical Trial to Explore the Drug Interaction of Tegoprazan or RAPA113 and Clopidogrel After Oral Administration in Healthy Male Volunteers
Brief Title: Effect of Tegoprazan or RAPA113 on Pharmacodynamics/Pharmacokinetics of Clopidogrel in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_APA_113
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel; tegoprazan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clopidogrel 75 mg (Active Comparator): Oral administration of clopidogrel 75 mg tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75mg
- Clopidogrel 75 mg + Tegoprazan 50 mg (Experimental): Oral administration of clopidogrel 75 mg tablet and Tegoprazan 50mg tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75mg; Drug: Tegoprazan 50 mg
- Clopidogrel 75 mg + RAPA113 (Experimental): Oral administration of clopidogrel 75 mg tablet and RAPA113 tablet once daily for 7 days
  Interventions: Drug: Clopidogrel 75mg; Drug: RAPA113

INTERVENTIONS:
Drug: Clopidogrel 75mg — Clopidogrel 75 mg tablet
  Other Names: Plavix
Drug: Tegoprazan 50 mg — Tegoprazan 50 mg tablet
  Other Names: K-CAB
  Arms: Clopidogrel 75 mg + Tegoprazan 50 mg
Drug: RAPA113 — RAPA113 tablet
  Arms: Clopidogrel 75 mg + RAPA113

SUMMARY:
This study aims to evaluate the influence of tegoprazan or RAPA113 on the pharmacodynamics/Pharmacokinetics of following co-administration of tegoprazan or RAPA113 and clopidogrel in healthy male volunteers.

DETAILED DESCRIPTION:
Evaluation Criteria:

* Primary outcome Pharmacodynamic assessments using P2Y12 assay
* Secondary outcome Pharmacokinetics assessments on Cmax,ss, AUCτ,ss, tmax,ss, Cmin,ss , CLss/F of Clopidogrel
* Safety assessments with adverse event monitoring including subjective/objective symptoms, physical examination, vital signs, electrocardiogram, and laboratory test

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged ≥ 19 years and ≤ 50 years on the date of the written informed consent
* Body weight of ≥ 55.0 kg and ≤ 90.0 kg, with body mass index (BMI) of ≥ 18.5 kg/m2 and ≤ 27.0 kg/m2 at the time of screening
* Helicobacter pylori negative
* Voluntarily decided to participate in the study and provided written informed consent before any screening procedure

Exclusion Criteria:

* Has a history of or currently has clinically significant liver, kidney, nervous system, immune system, respiratory system, endocrine system, blood, tumor, cardiovascular system or psychiatric disease
* Has a history of gastrointestinal diseases (such as Crohn's disease, ulcer, etc.) or surgery (except for simple appendectomy or hernia) that can affect the absorption of drugs
* Has a genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Has a clinically significant history of hemorrhage (e.g. Gastric ulcers, intracranial bleeding, haemophilia, gastrointestinal bleeding, urinary tract bleeding, vitreous hemorrhage, etc.)
* P2Y12 Reaction Unit (PRU) by P2Y12 assay outside the upper/lower limit of normal range by 10% at screening
* Considered ineligible to participate in the study based on screening test(by asking condition, vital sign, 12-lead ECG, physical exam, laboratory test etc.) results :

  1. Platelet, PT and aPTT levels outside the upper/lower limit of normal range by 10%
  2. AST (GOT), and ALT (GPT) levels greater than 1.25x of the upper limit of normal range
  3. Blood total bilirubin levels greater than 1.5x of the upper limit of normal range
  4. Hemoglobin levels less than 12.0 g/dL
  5. eGFR (estimated Glomerular Filtration Rate) using MDRD (Modification of Diet in Renal Disaster) < 60 mL/min/1.73 m2

     : eGFR (estimated glomerular filtration rate) (mL/min/1.73m2) = 175 x [serum creatinine (mg/dL)]-1.154 x [age]-0.203
  6. positive as a result of serum examination (B-type hepatitis test, hepatitis C test, human immunodeficiency virus test, syphilis test)
  7. Systolic blood pressure < 90 mmHg or > 150 mmHg, diastolic blood pressure < 50 mmHg or > 100 mmHg, or pulse rate < 45 beats/minute or > 100 beats/minute when vital signs are measured in sitting position after resting for at least 5 minutes during screening

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Change in P2Y12 Reaction Unit (PRU) from baseline | Pre-dose(0h) on days 1, 3, 5, 7 and 8 in each period
  Pharmacodynamics blood sampling to measure PRU using VerifyNow® system

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Principal Investigator — Severance Hospital, Dept of Clinical Pharmacology
Locations (1):
- Severance Hospital, Seoul, South Korea